CLINICAL TRIAL: NCT04867096
Title: Effects of a Supervised Exercise on Sleep in Patients With Non Metastatic Breast Cancer During Chemotherapy
Brief Title: Supervised Exercise, Sleep in Patients With Non Metastatic Breast Cancer
Acronym: FATSOMCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/482
Record Dates: First submitted 2021-04-16; First posted 2021-04-30 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity intervention (Experimental): Arm A : "standard oncologic care coupled with physical activity intervention (3 times / week) " during 3 months.
  Interventions: Other: Physical activity
- Control (No Intervention): Arm B : "standard oncologic care".

INTERVENTIONS:
Other: Physical activity — Patients in arm A (interventional) will carry out a physical activity intervention during 3 months. Patients should perform an interval training program on cycle-ergometer during 3 sessions per week.
  Arms: Physical activity intervention

SUMMARY:
Insomnia affects about 60% of the patients treated with radio-chemotherapy, a percentage twice higher compared to that observed in the general population. This sleep disorder increases cancer-related fatigue (CRF), the side effect most often reported by patients. Conversely, it is well accepted that adapted physical activity (APA) improves tolerance to treatment, decreases the risk of recurrence, increases survival, and reduces CRF. The present study aims to evaluate, in non-metastatic breast cancer patients, the composition and architecture of sleep by ambulatory polysomnography and to verify the effects of an APA rehabilitation program (3 times a week during 12 weeks), on the quality and quantity of sleep, daytime sleepiness. The biological markers: melatonin and body temperature will be studied to better understand the chronobiological mechanisms of the sleep-wake rhythm. Finally, the physiological responses to exercise, pain, CRF and finally quality of life will be studied at the beginning, at the end of the program and at a distance from it. Improved sleep-wake rhythm by a physical activity may reduce CRF, prevent recurrence and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65
* Patients with non-metastatic breast cancer undergoing chemotherapy
* Patients with insomnia
* Certificate of non-contraindication to the practice of physical activity
* Women who have been postmenopausal for at least 24 months, surgically sterilized, or, for women of childbearing potential, use an effective method of contraception (oral contraceptives, contraceptive injections, intrauterine devices, double-barrier method, contraceptive patches)
* Signature of informed consent to participate indicating that the subject has understood the purpose and procedures required by the study and that he agrees to participate in the study and to comply with the requirements and restrictions inherent in this study
* Affiliation to a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Patients treated with melatonin or taking hypnotics
* Patients with metastases
* Oxygen saturation at rest (SaO2) ≤ 92%
* Patients without insomnia and / or sleep disorders
* Autoimmune disease (systemic lupus erythematosus, rheumatoid arthritis)
* Symptomatic osteoarthritis, cardiovascular disease (angina pectoris or uncontrolled hypertension) or lung disease (chronic obstructive pulmonary disease)
* Patients suffering from malnutrition (BMI <18 kg.m-2) or weight loss> 10% during the previous 3 months
* Patients with psychiatric or cognitive disorders deemed unsuitable for physical activity
* Pregnant or breastfeeding women
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate with the study and / or weak cooperation anticipated by the investigator
* Subject without health insurance
* Subject being in the period of exclusion from another study or provided for by the "national file of volunteers".

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Total sleep time at 6 months | 6 months
  Evaluated with polysomnography

SECONDARY OUTCOMES:
Change from baseline quality of sleep at 6 months | 6 months
  Evaluated with actimetry
Change from baseline Score of fatigue at 6 months | 6 months
  Evaluated with questionnaire Multidimensional Fatigue Inventory (score between 20 to 100)
Change from baseline body composition at 3 months | 3 months.
  Evaluated bioimpedance BMI in Kg/m2
Score of pain | Baseline (T0) , 3 months (T3).
  Evaluated by questionnaire Brief Pain Inventory-Short Form (score between 15 to 150)
Inflammatory responses | Baseline (T0), 3 months (T3).
  Evaluated with enzyme-linked immunosorbent assay (ELISA)
Level of physical activity | Baseline (T0), 3 months (T3), 6 months (T6).
  Evaluated with smartwatch withings with number of step
Basic respiratory functional exploration | Baseline (T0), 3 months (T3).
  Evaluated by pneumotachography (Sensors Medics MSE, USA) for the evaluation of bronchial volumes and flows.
Level of anxiety | Baseline (T0), 3 months (T3), 6 months (T6).
  Evaluated by questionnaire Hospital Anxiety and Depression scale (under 7 to more than 11)
Concentration of Melatonin | Baseline (T0), 3 months (T3), 6 months (T6).
  Evaluated by saliva samples
Body temperature | Baseline (T0), 3 months (T3), 6 months (T6).
  Evaluated by thermobuttons

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drozd C, Curtit E, Jacquinot Q, Marquine C, Mansi L, Chaigneau L, Dobi E, Viot J, Meynard G, Paillard MJ, Goujon M, Roux P, Vernerey D, Gillet V, Bourdin H, Galli S, Meneveau N, Mougin F. A randomized trial to evaluate the effects of a supervised exercise program on insomnia in patients with non-metastatic breast cancer undergoing chemotherapy: design of the FATSOMCAN study. BMC Cancer. 2023 May 17;23(1):449. doi: 10.1186/s12885-023-10902-6. PMID 37198562